CLINICAL TRIAL: NCT00526227
Title: Clinical Study to Evaluate System Safety and Clinical Performance of the SecuraTM ICD
Brief Title: SecuraTM ICD Clinical Evaluation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Results first posted 2009-06-10 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2020-11

CONDITIONS: Tachyarrhythmias
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Secura ICD implant (Experimental): Secura ICD device implanted
  Interventions: Device: Secura ICD

INTERVENTIONS:
Device: Secura ICD — Secura Implantable Cardioverter Defibrillator (ICD) will be implanted
  Other Names: Secura TM

SUMMARY:
The purpose of the Secura clinical study is to evaluate the overall system safety and clinical performance of the Secura DR Implantable Cardioverter Defibrillator (ICD)

DETAILED DESCRIPTION:
The Secura ICD is an investigational dual chamber ICD that provides atrial and ventricular tachyarrhythmia detection and therapy, cardioversion, defibrillation, dual chamber rate-responsive bradycardia pacing and diagnostics.

The study will be a prospective, non-randomized, multicenter clinical study, conducted in approximately 15 centers.

To allow for sufficient experience with the device, a maximum of 80 subjects may be implanted with the Secura device. Data will be collected at baseline (enrollment), implant, 1-, 3-, and 6- months post implant and every 6 months thereafter or until study closure (whichever occurs first), Unscheduled Follow-up visits, System Modifications, Technical Observations, Study Deviations, Study Exit, upon notification of new or updated Adverse Events and in case of death.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have an ICD indication.
* Patients who are geographically stable and available for follow-up at the study center for the duration of the study.
* Patients who have signed a Medical Ethics Committee (MEC) approved Informed Consent form.

Exclusion Criteria:

* Patients with a life expectancy less than the duration of the study.
* Patients with medical conditions that preclude the testing required for all patients by the study protocol or that otherwise limit study participation required for all patients.
* Patients with mechanical tricuspid heart valves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Secura Clinical Study Team, Study Chair — Medtronic Cardiac Rhythm and Heart Failure
Locations (13):
- Wels, Austria
- Tampere, Finland
- Germany (6):
  - Goettigen
  - Hanover
  - Homburg/Saar
  - Kaiserslautern
  - Lüdenscheid
  - Münster
- Athens, Greece
- Netherlands (2):
  - Breda
  - Enschede
- Riyadh, Saudi Arabia
- Lund, Sweden

REFERENCES:
- [Derived] Murgatroyd FD, Helmling E, Lemke B, Eber B, Mewis C, van der Meer-Hensgens J, Chang Y, Khalameizer V, Katz A. Manual vs. automatic capture management in implantable cardioverter defibrillators and cardiac resynchronization therapy defibrillators. Europace. 2010 Jun;12(6):811-6. doi: 10.1093/europace/euq053. Epub 2010 Mar 14. PMID 20231152

RESULTS

PARTICIPANT FLOW:
Groups:
- Secura ICD Implant: Participants were implanted with a Secura Implantable Cardiac Defibrillator (ICD)
Period: Overall Study
Arm/Group | Secura ICD Implant
Started | 81
Completed | 79
Not Completed | 2
Not completed — Device not implanted | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: 80 participants were implanted with a Secura ICD, but the primary objective analysis was done on 44 participants.
Groups:
- Secura Implant: Patients implanted with Secura device
Arm/Group | Secura Implant
Number analyzed (Participants) | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (10.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 63
Region of Enrollment [Number; unit: participants]
  Austria | 10
  Germany | 48
  Netherlands | 10
  Greece | 4
  Saudi Arabia | 3
  Finland | 3
  Sweden | 3

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Unanticipated Serious Adverse Device Effects at 1-month Post Implant.
Description: Criteria to assess the results of the primary objective safety analysis is to demonstrate that the percentage of subjects experiencing an Unanticipated Serious Adverse Device Effect (USADE) is lower than 10% at one-month post-implant, with one month considered to be the same as 28 days.
  A pre-specified interim analysis is included in the study which, if the primary objective was met, is to also be considered the final analysis.
Time Frame: 1 month
Population: Forty-four (44) out of the 80 subjects completed at least one-month (28 days) of follow-up post-implant and were included in the (interim) analysis for the primary objective. One subject of the 80 implanted subjects died prior to the 1-month follow-up.
Measure: Number (97.5% Confidence Interval); unit: percentage of patients
Groups:
- Secura Implant: Patients implanted with a Secura device
Arm/Group | Secura Implant
Number analyzed (Participants) | 44
percentage of patients | 0 [0 to 7.7]
Statistical Analysis 1: Comparison: Secura Implant; H 0 (null hypothesis): P ≥ 10%; H A (alternative hypothesis): P < 10%, where P is the percentage of subjects experiencing a USADE through the 1-month post implant. An upper limit of the confidence interval of the percentage subjects with USADE not greater than or equal to 10% at the 1-month follow-up visit provides a reasonably-sized clinical study with sufficient power to detect USADEs; Test type: Other — An exact one-sided 97% upper confidence bound or a p-value will be calculated based on the observed percentage of subjects with an USADE within the first month post-implant. This rate will be considered acceptable if the one-sided 97% upper confidence bound is less than 10% or, equivalently, if the p-value is less than 0.0304; Percentage = 7.7 — The CI was calculated based on 44 patients at interim analysis: 0 USADE were reported within 1-month post implant, ie 0% of subjects experienced a USADE. The one-sided 97% exact binomial upper confidence bound was 7.7% which is lower than 10%

2. Secondary Outcome: System Performance Assessed by Holter Records
Description: The first 21 digital Holter records that were successfully collected in the total of 80 implanted participants will summarize any anomalous or unintended operation and describe device features, ventricular arrhythmia detection times and device classification of ventricular arrhythmias.
Time Frame: 1 month
Population: All implanted participants underwent Holter recording. The first 21 Holter recordings that were successful were analyzed.
Measure: Number; unit: anomalous or unintended operation
Units Other Than Participants: Holter recordings
Groups:
- Secura Implant: The first 21 patients implanted with a Secura device that has a successful Holter recording
Arm/Group | Secura Implant
Number analyzed (Participants) | 21
Number analyzed (Holter recordings) | 21
anomalous or unintended operation | 0

3. Secondary Outcome: Adverse Events
Description: Number of Adverse Events reported in the implanted subjects.
Time Frame: 1 Month
Measure: Number; unit: adverse events
Arm/Group | Secura Implant
Number analyzed (Participants) | 79
adverse events | 62

4. Secondary Outcome: System Performance Assessed by Save to Disk Files
Description: The Save to Disk files from 79 implanted participants collected after implant and 1 month follow up were reviewed to identify any anomolous or unintended device operation, examine device features, observe ventricular arrhythmia detection times and device classification of ventricular arrhythmias.
Time Frame: 1 month follow-up
Population: Save to Disk files were collected for all participants implanted with a Secura ICD after implant and 1 month follow up.
Measure: Number; unit: anomolous or unintended device operation
Groups:
- Secura ICD Implant: Participants were implanted with a Secura ICD
Arm/Group | Secura ICD Implant
Number analyzed (Participants) | 79
anomolous or unintended device operation | 0

5. Secondary Outcome: System Performance Assessed by Technical Observations
Description: Reported technical observations will be reviewed to determine if there are any device performance issues.
Time Frame: 1 month follow-up
Population: One (1) technical observation was reported in the 79 participants that were implanted with a Secura ICD.
Measure: Number; unit: device performance issues
Units Other Than Participants: Reported Technical Observations
Arm/Group | Secura ICD Implant
Number analyzed (Participants) | 1
Number analyzed (Reported Technical Observations) | 1
device performance issues | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, contracts allow investigators to publish study results per the publication plan/protocol following Medtronic's review to determine whether Confidential Information (CI) is disclosed. Any such CI is deleted prior to publication/presentation. Medtronic may not censor/interfere with the publication except as described. Investigators may not publish any single-site publications until the main multi-site study publication has occurred.